CLINICAL TRIAL: NCT06620744
Title: Magnetocardiography (MCG) Device Use in Patients With Elevated Troponin
Acronym: DUET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SB Technology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SB-ACS-004
Record Dates: First submitted 2024-09-20; First posted 2024-10-01 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2024-09

CONDITIONS: ACS - Acute Coronary Syndrome
Keywords: magnetocardiography; MCG
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Sponsor MCG Device (Experimental): All participants will receive a scan from the sponsor's MCG device.
  Interventions: Device: Sponsor MCG deivce

INTERVENTIONS:
Device: Sponsor MCG deivce — Unshielded device measuring cardiac magnetic fields.

SUMMARY:
This prospective device study will examine the feasibility of MCG data collection in a hospital setting using the SandboxAQ MCG device as a potential method to more accurately and quickly quantify cardiac disease of patients with elevated Troponin.

ELIGIBILITY:
Inclusion Criteria:

* Received a positive hs-cTnI based on the institutions laboratory normal value ranges (e.g. female ≥14 and male ≥35)

Exclusion Criteria:

* Present STEMI
* Having an active atrial fibrillation episode as seen on 12-lead ECG
* Clear non-ischemic cause for symptoms (e.g. trauma)
* Active thoracic metal implants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-09-21 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Proportion (%) of all collected MCG data that meets the necessary data quality. requirements and are deemed suitable for analysis. | Per-scan, on average 5 minutes, day of enrollment
  MCG Data Quality

SECONDARY OUTCOMES:
Sandbox MCG safety | 30-days
  Device-related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Kit Yee Au-Yeung, PhD, Study Director — SB Technology, Inc.
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No